CLINICAL TRIAL: NCT02865694
Title: Developing and Implementing Familial Hypercholesterolemia Registry in Isfahan, Iran: Cascade Screening, Management and Long-term Follow up.
Brief Title: Developing and Implementing Familial Hypercholesterolemia Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohamamd Reza Sabri, Head of Pediatric Cardio vascular research Center, Isfahan University of Medical Sciences
Other Study IDs: FH-ICRI
Record Dates: First submitted 2016-08-10; First posted 2016-08-12 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Plasma, buffy coat, blood.

INTERVENTIONS:
Other: Cascade

SUMMARY:
Familial hypercholesterolemia (FH) is a most prevalent genetic disorder define as high cholesterol level and premature death. The prevalence of FH reported in few countries however unknown in Iran. Thus determine the FH patient, finding diagnostic strategy and appropriate treatment are important. We intent to use cascade method to screening patients, also our expected outputs are to develop and implement a registry program for FH patients and their families and to study their genetic disorder. FH patients will be followed from management, treatment and prevention of Cardio vascular disease in order to increase premature death.

DETAILED DESCRIPTION:
Familial hypercholesterolemia (FH) is a genetic disorder define as high cholesterol levels, particularly very high levels of low-density lipoprotein (LDL), in the blood and early cardiovascular disease and premature death. FH is an autosomal dominant disease with a prevalence 1:500 (new study in Netherlands demonstrated 1:244) in population more frequent than Cystic fibrosis, mellitus diabetes or neonatal hypothyroidism. Canadian registry demonstrated FH is more common among people if French Canadian, Christian Lebanese, and Afrikaner descent. The Major causes of FH are pathogenic variant in the LDL-receptor (LDLR) gene or the Apo lipoprotein B (APOB) gene. The clinical signs of FH are high level of Cholesterol (between 350-550 mg/dL in heterozygous), Yellow deposits of cholesterol-rich fat in various places on the body such as around the eyelids (known as xanthelasma palpebrarum), the outer margin of the iris (known as arcus senilis corneae), and in the tendons of the hands, elbows, knees and feet, particularly the Achilles tendon (known as a tendon xanthoma). FH is a hidden syndrome which leads to cardiovascular disease.

After introducing the statins total mortality have reduced significantly in these patients. Thus screening and identification of patients and treatment with the most effective therapies will decrease the risk of premature death.

Also, most of patients require an appropriate lipid-lowering medications. Although the genetic problem is the most important factor to expression of FH other factors like environmental and metabolic factor can be effective in CVD and premature death.

Therefore, identification and follow-up FH patients is important for CVD Rate cuts and decrease Treatment costs thus this study can gain these outcomes.

ELIGIBILITY:
Inclusion Criteria:

Personal concentration of LDL-C > 190 mg/dL or LDL-C > 120 mg/dL in Treatment Group.

Family and/or personal history of premature heart disease.

Exclusion Criteria:

Hyperlipidemia with underlying disorders.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from clinical laboratory.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with FH. | 1 Year

SECONDARY OUTCOMES:
Number of premature cardio vascular events annually follow-up. | 5 Years
Low Density Lipoprotein (LDL-C) at base line and during annually follow-up. | 1 Year
High density lipoprotein (HDL) at base line and during annually follow-up. | 1 Year
triglyceride (TG) at base line and during annually follow-up. | 1 Year
LDL-receptor frequency of mutation in Persian population. | 1 Year
PCSK9 frequency of mutation in Persian population. | 1 Year
Apo-B frequency of mutation in Persian population. | 1 Year

CONTACTS AND LOCATIONS:
Locations (1):
- Isfahan Cardio vascular Research Institute, Isfahan, Iran